CLINICAL TRIAL: NCT02536352
Title: Effect of Supplementation of Fluoride on Maternal Periodontal Health, Preterm Delivery, and Perinatal Well-Being
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: IRB00038838
Record Dates: First submitted 2015-08-27; First posted 2015-08-31 (Estimated); Last update posted 2019-11-05 (Actual); Status verified 2019-11

CONDITIONS: Preterm Birth; Preterm Labor; Bacteremia; Preterm Premature Rupture of Fetal Membranes
Keywords: Fluoride Supplementation; Prenatal Vitamin; Pregnancy Nutrition; Prenatal Nutrition
MeSH Terms: conditions — Premature Birth; Obstetric Labor, Premature; Bacteremia; Fetal Membranes, Premature Rupture | interventions — Fluorides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fluoride prenatal vitamin (Experimental): Prenatal vitamin-mineral containing 3 mg fluoride
  Interventions: Drug: Prenatal vitamin-mineral containing 3 mg fluoride
- Standard prenatal vitamin (Active Comparator): Prenatal vitamin-mineral containing 0 mg fluoride
  Interventions: Dietary Supplement: Prenatal vitamin-mineral containing 0 mg fluoride

INTERVENTIONS:
Drug: Prenatal vitamin-mineral containing 3 mg fluoride — Prenatal vitamin-mineral containing 3 mg fluoride to be taken daily, starting at 10-20 weeks gestation until delivery.
  Arms: Fluoride prenatal vitamin
Dietary Supplement: Prenatal vitamin-mineral containing 0 mg fluoride — Prenatal vitamin-mineral containing 0 mg fluoride to be taken daily, starting at 10-20 weeks gestation until delivery.
  Arms: Standard prenatal vitamin

SUMMARY:
The purpose of this study is to determine whether fluoride supplementation during pregnancy is effective in extending the length of gestation and improving overall perinatal well-being.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention (CDC) reports that preterm birth affected about 1 in 10 infants born in the United States in 2015. These statistics emphasize the significance of implementing a safe and effective therapy into routine clinical care aimed at reducing the rate of preterm birth. There has been evidence to suggest that fluoride supplementation to women during pregnancy can provide other medical benefits, in addition to a reduction in dental caries.

Fluoride is recognized by the Food and Nutrition Board (F&NB) of the American Academy of Sciences and the Food & Drug Administration (FDA) as an essential ion due to its association with a reduction in dental caries.

Upon entering the body, fluoride is taken up into the bones/calcified tissues, and excreted by the kidneys. When supplied during pregnancy in small aliquots, as with water fluoridation, the fluoride is likely taken up in the mother's bones and excreted by her kidneys so rapidly, that the fetus is denied a meaningful amount of fluoride, unless it is supplied in a pulse dose by supplement. The Institute of Medicine's Food and Nutrition Board recommends 3 mg/day for Adequate Intake in pregnancy and deems 10 mg/day as the Upper Limit.

After several papers elucidating an association between poor dentition, periodontal disease, and preterm birth, subsequent RCT's of regular periodontal scaling and treatment during pregnancy are still inconclusive in regards to preterm birth.

The investigators hypothesize that fluoride supplementation during pregnancy may have a beneficial effect on the natural microbiome of the maternal oral cavity and genital tract, capable of protecting against transient bacteremia and ascending infection, respectively, which are known antecedents to both preterm labor and preterm premature rupture of membranes. The research team predicts that the testing and analysis of specimens collected will demonstrate microbiome changes toward a more favorable profile not associated with preterm birth.

The proposed randomized, double-blinded, placebo-controlled clinical trial aims to confirm the efficacy of fluoride supplementation in pregnancy to extend length of gestation and increase overall perinatal well-being, and to confirm transplacental transfer of supplemental fluoride. This research may also identify other beneficial maternal and neonatal outcomes associated with the administration of fluoride during the perinatal period by attempting to characterize and compare the microbiomes of the maternal oral cavity and genital tracts between supplemented and unsupplemented gravidas.

ELIGIBILITY:
Inclusion Criteria:

* Women who are between 10-20 weeks gestational age at the time of recruitment
* Delivery at Johns Hopkins Hospital or Johns Hopkins Bayview Medical Center

Exclusion Criteria:

* Use of prescription strength, high dose fluoride products (greater than 0.76% of fluoride), prescribed by a dental professional (toothpastes, mouthwashes, topical treatments). All over-the-counter toothpaste and mouthwash products are acceptable to use.
* Occupational exposure to fluoride.
* The daily amount of fluoride ingested should not exceed 10 mg/day, according to the Institute of Medicine and the FDA. Any participants consuming amounts of fluoride close to 10 mg/day will be excluded.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2015-10; Primary Completion 2019-10-01 (Actual); Study Completion 2019-10-01 (Actual)

PRIMARY OUTCOMES:
Length of gestation | Participants will be followed from the time of study enrollment until delivery, up to 30 weeks total in the study
  the length of gestation will be measured in weeks at time of delivery

SECONDARY OUTCOMES:
Birth weight | Participants will be followed from the time of study enrollment until delivery, up to 30 weeks total in the study
  Birth weight will be measured in grams and pounds
Birth length | Participants will be followed from the time of study enrollment until delivery, up to 30 weeks total in the study
  birth length will be measured in inches
Preterm birth | Participants will be followed from the time of study enrollment until delivery, up to 30 weeks total in the study
  Preterm birth will be measured in weeks at time of delivery
Preterm premature rupture of membranes (PPROM) | Participants will be followed from the time of study enrollment until delivery, up to 30 weeks total in the study
  PPROM will be measured in weeks at time of PPROM

CONTACTS AND LOCATIONS:
Overall Officials: Irina Burd, M.D., Ph.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

REFERENCES:
- [Background] Leverett DH, Adair SM, Vaughan BW, Proskin HM, Moss ME. Randomized clinical trial of the effect of prenatal fluoride supplements in preventing dental caries. Caries Res. 1997;31(3):174-9. doi: 10.1159/000262394. PMID 9165186
- [Background] Srinivas SK, Sammel MD, Stamilio DM, Clothier B, Jeffcoat MK, Parry S, Macones GA, Elovitz MA, Metlay J. Periodontal disease and adverse pregnancy outcomes: is there an association? Am J Obstet Gynecol. 2009 May;200(5):497.e1-8. doi: 10.1016/j.ajog.2009.03.003. PMID 19375568
- [Background] Institute of Medicine (US) Standing Committee on the Scientific Evaluation of Dietary Reference Intakes. Dietary Reference Intakes for Calcium, Phosphorus, Magnesium, Vitamin D, and Fluoride. Washington (DC): National Academies Press (US); 1997. Available from http://www.ncbi.nlm.nih.gov/books/NBK109825/ PMID 23115811
- [Background] Iheozor-Ejiofor Z, Middleton P, Esposito M, Glenny AM. Treating periodontal disease for preventing adverse birth outcomes in pregnant women. Cochrane Database Syst Rev. 2017 Jun 12;6(6):CD005297. doi: 10.1002/14651858.CD005297.pub3. PMID 28605006